CLINICAL TRIAL: NCT04928872
Title: The Relation Between the Meal Macronutrient Distribution and Plasma Metabolites to Model the Composition of Meals of Patients With Diabetes II and Cardiovascular Disease.
Brief Title: Macronutrient Distribution and Plasma Metabolites to Model Meals Composition
Status: Completed | Type: Observational
Sponsor: Texas A&M University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Professor & Chancellor Edges Fellow, Texas A&M University
Other Study IDs: 2017-0886
Record Dates: First submitted 2021-06-01; First posted 2021-06-16 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Glucose Metabolism
Keywords: response to food; plasma glucose; continuous glucose monitor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-diabetic older adults: Non-diabetic older adults
  Interventions: Combination Product: Predefined meal

INTERVENTIONS:
Combination Product: Predefined meal — Nine predefined meals are administered in a randomized fashion, one meal per one study day, 2-3 study days per week. Meals have a form of drinks with different compositions of protein, carbohydrates and fat in relation to the US diet

SUMMARY:
Continuous glucose monitors (CGMs) measure plasma glucose concentration continually and thus they are a key tool in the management of diabetes, including type 2 diabetes (T2D). A key factor in diabetes management is a reduction of dietary carbohydrates (CHO) and/or exchanging high glycemic index (GI) CHO with low GI CHO. However, the protein and fat content of the meal can have a significant impact on the glucose readings obtained from a CGM as there is no enough data available on their sensitivity during meals.

DETAILED DESCRIPTION:
The study involves 1 screening visit of approximately 1 hour and 9 study days of approximately 8 hours. Subjects will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight, height, and body composition by Dual-energy X-ray absorptiometry (DXA) will be measured. In addition, habitual dietary intake, physical activity level (PASE), and quality of life (SGRQ-C) will be assessed.

To test the relation between plasma amino acid, triglycerides, and glucose concentration measured by standard methods (such as finger stick) and continuous wearable devices, a premarket FDA-approved continuous glucose monitor (CGM) from Abbott (FreeStyle Libre Pro) that monitors glucose concentrations every 15 min is used. The single-use sensors are placed on the upper arm and contain a very tiny 5 mm filament (<0.4 mm diameter) that is introduced into the skin when the sensor is placed. On the first study day, the CGM will be placed to monitor glucose concentrations until the last study day. At least every 14 days, sensors will be replaced by new ones. On each study day, body weight and height will be measured and the glucose concentration data will be downloaded from the sensor onto the reader device. A catheter will be inserted in a peripheral vein of the lower arm or hand to enable blood sampling. The arm will be put in a hot box to allow collecting arterialized venous blood samples. After taking a baseline blood sample, the predefined meal will be consumed within 10 min. Small arterialized venous blood samples (5 ml) will subsequently be drawn at times: 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 420, and 480 minutes (13 blood samples, total blood approx 65 ml). Samples will be collected in predefined tubes, plasma/serum separated, aliquoted, and stored at -80 deg. Celsius for later assays and/or send to a local accredited laboratory for the concentrations of amino acids and other parameters (including fatty acids, glucose, insulin).

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk, sit down and stand up independently
* Ability to lie in a supine or slightly elevated position for 8.5 hours
* BMI between 25 and 35 kg/m2
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Established diagnosis of malignancy
* Established diagnosis of Insulin-Dependent Diabetes Mellitus
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults (60-85y; equal gender) with a BMI between 25 and 35 will be recruited from an existing database of CTRAL. In addition, we will recruit older adults that respond to distributed flyers and advertisements in the newspaper and to radio announcements in the community of the College Station/Bryan area. Informed consent will be obtained on the screening day before any study-related procedures will be performed. If inclusion/exclusion criteria are met, subjects are invited to take part in the study.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Prediction models of postprandial plasma amino acid patterns in relation to the macronutrient content of predefined meals as assessed by plasma concentrations of amino acids, glucose, and/or triglycerides | 9 study visits: one meal per one study day, 2-3 meals per week, 8-hour blood blood sample collection after a meal intake. Study completion: 4-5 weeks.
  Participants consume 9 predefined meals in the fasted state with macronutrient composition reflecting common meals in the US diet. One meal is consumed during one study visit with a total of 9 visits. A baseline sample is collected followed by an intake of one meal during one study visit. Blood samples (in the 15-and 30-minutes interval) are collected for 8 hours after a meal intake. Collected plasma will be used for amino acid analysis. Statistical models will be used to predict plasma amino acids from patterns of amino acids, glucose, and/or triglycerides in the consumed meals.

SECONDARY OUTCOMES:
Discordance of glucose measurement after an intake of the predefined meal as measured by a fingerstick, continuous glucose monitor, and certified laboratory | 9 study visits: one meal per one study day, 2-3 meals per week, 8-hour blood blood sample collection after a meal intake. Study completion: 4-5 weeks.
  A continuous glucose monitor is placed during the first study visit. Participants consume 9 predefined meals in the fasted state with macronutrient composition reflecting common meals in the US diet. One meal is consumed during one study visit. A baseline sample is collected followed by an intake of one meal during one study visit. Blood samples (in the 15-and 30-minutes interval) for glucose measurements are taken and plasma samples are collected. Plasma glucose is measured by a glucose monitor and outsourced to the certified laboratory. Information from continuous glucose monitor is collected at the end of each study day.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas EP Deutz, MD, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barua S, A Wierzchowska-McNew R, Deutz NEP, Sabharwal A. Discordance between postprandial plasma glucose measurement and continuous glucose monitoring. Am J Clin Nutr. 2022 Oct 6;116(4):1059-1069. doi: 10.1093/ajcn/nqac181. PMID 35776949